CLINICAL TRIAL: NCT03456115
Title: Assessing Mechanical Nasal Obstruction, a Potential New Treatment Option.
Brief Title: A New Treatment for Mechanical Nasal Obstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00135539
Record Dates: First submitted 2018-02-13; First posted 2018-03-07 (Actual); Results first posted 2023-07-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-06

CONDITIONS: Nasal Obstruction
Keywords: nasal obstruction; nasal valve collapse
MeSH Terms: conditions — Nasal Obstruction

STUDY DESIGN:
Intervention Model Description: All participants will undergo the same intervention, which is a trial of various internal nasal dilators.
Masking Description: Participants will be unaware of which nasal dilator they are trialing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Mechanical Nasal Dilator (Experimental): All participants will be trialing the 5 devices and reporting their thoughts on comfort, and perception of symptoms of mechanical nasal obstruction by way of survey completion. The devices include 4 commercially available nasal dilators: Breathe Right, Max Air, Sleep Right, Nozovent, and the study team's investigational device dubbed the Schnozzle.
  Interventions: Device: Mechanical nasal dilator

INTERVENTIONS:
Device: Mechanical nasal dilator — Participants will be asked to trial 5 different mechanical nasal dilators. 4 of which are commercially available and one of which is the investigational device being studied for feasibility. The 4 commercially available nasal dilators include Breathe Right, Max Air, Sleep Right, Nozovent. The fifth device is the study team's investigational device dubbed the Schnozzle.

SUMMARY:
The research team has developed a prototype for an investigational mechanical nasal dilator and the investigators aim to evaluate its efficacy.

Specifically, the investigators wish to address the following research questions: 1) How does mechanical nasal obstruction affect patients' lives? The investigators aim to answer this question with use of validated questionnaires. 2) How do currently available mechanical nasal dilators affect objective and subjective findings related to nasal obstruction? This will be evaluated with objective nasal airflow testing and with modifications to validated questionnaires 3) How does the investigational team's novel device affect these same outcome measures? 4) Do patients find the investigational device subjectively comfortable and efficient?

DETAILED DESCRIPTION:
Background:

Restricted nasal breathing is a common complaint among patients presenting to Otolaryngology clinics. In fact, one in eight people experiences some degree of nasal obstruction, or regular difficulty breathing through the nose, which is often the result of a narrowing or collapse of the internal nasal valve. This condition is a daily source of discomfort that reduces productivity and quality of life. Sufferers report shortness of breath throughout the day, difficulty sleeping and habitual snoring, and limited stamina during sports and exercise.

Slight dilation of the nasal passages directly counteracts nasal obstruction and reverses symptoms in 89% of those afflicted. To this end, many patients undergo functional rhinoplasty procedures to surgically widen the nasal passages. However, up to 20% of patients experience unimproved or worsened symptoms postoperatively. Moreover, these surgeries are invasive, requiring autologous grafts taken from the nose, ear, or ribs; and surgeries entail a yearlong recovery period.

Nasal dilators such as Breathe Right strips offer a potential alternative to surgery, as these dilators mechanically expand the nasal passages to effectively relieve obstruction. However, existing products are designed as sleep aids, and customers find them uncomfortable, difficult to use, and too visible to wear in public. Although the mechanism for reversing nasal obstruction is straightforward, surgery is considered the only viable option for those who struggle to breathe during the day.

Engineers from the Johns Hopkins Biomedical Engineering Department, partnered with clinicians from the Johns Hopkins Department of Otolaryngology - Head and Neck Surgery, have developed the Schnozzle, a small silicone stent to counteract nasal valve collapse and relieve restricted nasal breathing. The investigators hypothesize that this device will improve symptoms of nasal obstruction and provide patients with a viable alternative to visible non-invasive devices or surgical management. The aim of this study is to evaluate the feasibility and comfort of this device in comparison to existing commercially available devices.

Recruitment:

Participants will be recruited from patients presenting to Otolaryngology clinics with symptoms of nasal obstruction. The otolaryngologist in clinic will screen these patients for nasal valve collapse as in standard clinical practice. This involves visualizing the nasal cavity through nasal endoscopy and evaluating the nasal valve using Cottle maneuver (applying lateral force to the cheek to open the nasal valve) or the modified Cottle maneuver (using a cotton tip applicator to open the nasal valve from inside the nasal cavity) and evaluating for improvement in nasal obstruction symptoms. Improved nasal airflow during the maneuver suggests nasal valve collapse contributes to restricted nasal airflow.

The clinical Otolaryngologist will counsel participants with nasal valve collapse regarding the various treatment options as in routine clinical practice (management options include to doing nothing, using existing nasal dilator devices, or undergoing surgery). Patients will then be invited to participate in the study, which will involve a study session in which patients are fitted with several nasal dilator devices, instructed in proper care and use, and report on their function and comfort. Additional participants will be recruited from patients who present to clinics with symptoms unrelated to nasal breathing to serve as a control group.

Study design:

If a patient expresses interest in participating, the patient will be introduced to a member of the research team to discuss the study and complete informed consent. All participation is voluntary and participants are able to withdraw from the study at any point. The study participant will be asked to complete a questionnaire, which includes the previously validated Nasal Obstruction and Septoplasty Effectiveness (NOSE) instrument, questions regarding the patient's current treatments, and a ranking of their preferred characteristics of an ideal nasal dilator.

Patients will then be asked to inhale rapidly into an airflow transducer to measure peak nasal inspiratory flow (PNIF). Following the pre-test survey participants will be fitted with existing nasal dilator products per manufacturer recommendations (Breathe Right strips, Max Air nose cones, Sleep Right dilator, and Nozovent dilator), and the experimental nasal dilators designed by the research team. In this crossover design study participants will be blinded as to which dilators are branded and which are experimental. The order of fitting nasal dilators will be randomized.

After each fitting and use for 5 minutes to adjust to the device and confirm there is no immediate discomfort or irritation, participants will undergo repeat PNIF testing with each device, then will be free to go home and trial the devices. Participants will be given a schedule specifying one device to use for at least one continuous hour per day in a randomized order, while also being blinded as to which device participants will be using (Schnozzle, Breathe Right, Max Air, Sleep Right, Nozovent). The devices will be numbered in a random fashion, for participants to be able to identify which device via the assigned number the devices are scheduled to use. Participants will similarly use the device number when performing any device evaluation. Participants are free to wear the assigned nasal dilator at their leisure, but must log the hours and activities performed while wearing the device (for example, "10am-11am exercising"). Participants are not required to wear a device in public at work or during exercise unless participants feel comfortable doing so. All devices should be worn overnight. If there is any discomfort, irritation, skin breakdown, or epistaxis the participant should stop wearing the device and contact the research team immediately. Each morning, the participant will complete a survey summarizing their experience using the assigned device. Before returning to the clinic for the conclusion of the study, participants may have several days without an assigned device. Participants are free to stop wearing all devices or use any device as participants please as long as it is consistent with proper care and use of the device(s).

After at least five days (one day per device) the participant will return to the office for an exit interview with the study team in regards to their subjective experience with each device. At the end of each trial participants will be asked to fill out a concluding survey regarding the device participants were using. At their exit interview participants will be asked to hand in the survey for each device participants trialed.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have presented to Otolaryngology clinics with complaints of nasal obstruction.
* Patients who have been found to have nasal valve collapse by an Otolaryngologist based on performance of the Cottle maneuver will be invited to participate in the study.
* Patients without evidence of nasal valve collapse, but are willing to participate in the study.

Exclusion Criteria:

* History of granulomatosis with polyangiitis, extensive prior sinus or turbinate surgery altering nasal cavity anatomy, pre-existing nasal mucosal injuries or abnormalities

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2022-05-12 (Actual); Study Completion 2022-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Rowan, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jessen M, Malm L. Definition, prevalence and development of nasal obstruction. Allergy. 1997;52(40 Suppl):3-6. doi: 10.1111/j.1398-9995.1997.tb04876.x. No abstract available. PMID 9353553
- [Background] Bloching MB. Disorders of the nasal valve area. GMS Curr Top Otorhinolaryngol Head Neck Surg. 2007;6:Doc07. Epub 2008 Mar 14. PMID 22073083
- [Background] Miman MC, Deliktas H, Ozturan O, Toplu Y, Akarcay M. Internal nasal valve: revisited with objective facts. Otolaryngol Head Neck Surg. 2006 Jan;134(1):41-7. doi: 10.1016/j.otohns.2005.08.027. PMID 16399179
- [Background] Camacho M, Zaghi S, Certal V, Abdullatif J, Modi R, Sridhara S, Tolisano AM, Chang ET, Cable BB, Capasso R. Predictors of Nasal Obstruction: Quantification and Assessment Using Multiple Grading Scales. Plast Surg Int. 2016;2016:6945297. doi: 10.1155/2016/6945297. Epub 2016 May 16. PMID 27293885
- [Background] Khosh MM, Jen A, Honrado C, Pearlman SJ. Nasal valve reconstruction: experience in 53 consecutive patients. Arch Facial Plast Surg. 2004 May-Jun;6(3):167-71. doi: 10.1001/archfaci.6.3.167. PMID 15148124
- [Background] Kiyohara N, Badger C, Tjoa T, Wong B. A Comparison of Over-the-Counter Mechanical Nasal Dilators: A Systematic Review. JAMA Facial Plast Surg. 2016 Sep 1;18(5):385-9. doi: 10.1001/jamafacial.2016.0291. PMID 27367589
- [Background] Picavet VA, Grietens J, Jorissen M, Hellings PW. Rhinoplasty from a rhinologist's perspective: need for recognition of associated sinonasal conditions. Am J Rhinol Allergy. 2012 Nov-Dec;26(6):493-6. doi: 10.2500/ajra.2012.26.3816. PMID 23232202
- [Background] Samaha M, Rassouli A. Spreader graft placement in endonasal rhinoplasty: Technique and a review of 100 cases. Plast Surg (Oakv). 2015 Winter;23(4):252-4. doi: 10.4172/plastic-surgery.1000944. PMID 26665141
- [Background] Kimbell JS, Frank-Ito DO. Mechanical Nasal Dilators for the Management of Nasal Obstruction. JAMA Facial Plast Surg. 2016 Sep 1;18(5):389-90. doi: 10.1001/jamafacial.2016.0656. No abstract available. PMID 27367256
- [Background] Raudenbush B. Stenting the nasal airway for maximizing inspiratory airflow: internal Max-Air Nose Cones versus external Breathe Right strip. Am J Rhinol Allergy. 2011 Jul-Aug;25(4):249-51. doi: 10.2500/ajra.2011.25.3621. PMID 21819762

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: All participants will be trialing the 5 devices and reporting their thoughts on comfort, and perception of symptoms of mechanical nasal obstruction by way of survey completion. The devices include 4 commercially available nasal dilators: Breathe Right, Max Air, Sleep Right, Nozovent, and the study team's investigational device dubbed the Schnozzle.
Period: Overall Study
Arm/Group | All Participants
Started | 36
Completed | 36
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Mechanical Nasal Dilator
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 29
  >=65 years | 6
Age, Continuous [Median (Full Range); unit: years] | 52 [17 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 15
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Change in Peak Nasal Inspiratory Flow (PNIF)
Description: PNIF will be measured using a PNIF meter. PNIF will be measured without any device in place and once during the fitting of each device. Flow is measured in liters per minute. Minimum value of -50, maximum value of 150 with higher scores indicating improved airflow.
Time Frame: Prior to device and after fitting each device (Up to 5 minutes)
Population: Same participants are showed in all arms because they received all interventions.
Measure: Mean (Standard Deviation); unit: liters per minute
Groups:
- Breathe Right: Breathe Right dilator
- Max Air: Max Air nose cones
- Sleep Right: Sleep Right dilator
- Mute: Mute dilator
- Nozovent: Nozovent dilator
- Schnozzle: Schnozzle dilator aka Hale
Arm/Group | Breathe Right | Max Air | Sleep Right | Mute | Nozovent | Schnozzle
Number analyzed (Participants) | 36 | 36 | 36 | 36 | 36 | 36
liters per minute | 28 (42) | 24 (38) | 13 (20) | 27 (47) | 25 (35) | 29 (40)

2. Secondary Outcome: Change in Nasal Obstruction and Septoplasty Effectiveness Scale (NOSE)
Description: The Nasal Obstruction and Septoplasty Effectiveness Scale (NOSE) aims to quantify symptoms of mechanical nasal obstruction. The NOSE metric has a scoring range go 0-100 with 0 being no symptoms of mechanical nasal obstruction and 100 being severe nasal obstruction.
  Each device is trialed for one day, hence the scale will be administered at Baseline and after a 24-hour trial of each of the 5 devices.
Time Frame: Baseline
Population: Nasal Obstruction and Septoplasty Effectiveness Scale (NOSE) was not captured on patients. Data was not collected.
Arm/Group | All Participants
Number analyzed (Participants) | 0

3. Secondary Outcome: Change in Nasal Obstruction and Septoplasty Effectiveness Scale (NOSE)
Description: as for outcome 2
Time Frame: 24-hour after trial of each device
Population: Nasal Obstruction and Septoplasty Effectiveness Scale (NOSE) was not captured on patients. Data was not collected.
Arm/Group | All Participants
Number analyzed (Participants) | 0

4. Secondary Outcome: Device Preference
Description: Participants will be asked to rank their preferred device form 1 (most preferred) to 5 (least preferred). The mean will be reported. Scores range from 1-5, with 1 being the most preferred.
Time Frame: Up to 5 days
Population: Same participants are showed in all arms because they received all interventions.
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Breathe Rite: Breathe Rite strips
- Nozovent Dilator: Nozovent dilator
  Participants will be asked to rank their preferred device form 1 (most preferred) to 5 (least preferred). The mean will be reported. Scores range from 1-5, with 1 being the most preferred.
- Schnozzle: Schnozzle dilator (aka Hale).
Arm/Group | Breathe Rite | Max Air | Sleep Right | Mute | Nozovent Dilator | Schnozzle
Number analyzed (Participants) | 36 | 36 | 36 | 36 | 36 | 36
score on a scale | 2.9 [1 to 5] | 5 [2 to 5] | 3.8 [1 to 5] | 2.7 [1 to 4] | 2.8 [1 to 4] | 3.8 [1 to 4]

ADVERSE EVENTS:
Time Frame: Data were collected during device use over a period of 5 days.
Description: Same participants are showed in all arms because they received all interventions.
Groups:
- Breathe Right: Breathe Right strips
Arm/Group | Breathe Right | Max Air | Sleep Right | Mute | Nozovent | Schnozzle
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/36 | 0/36 | 0/36 | 0/36 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36 | 0/36 | 0/36 | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 0/36 | 0/36 | 0/36 | 0/36 | 0/36 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-07-06): https://cdn.clinicaltrials.gov/large-docs/15/NCT03456115/Prot_SAP_ICF_000.pdf